CLINICAL TRIAL: NCT05999630
Title: The Use of Artificial Tears to Prevent Nasolacrimal Duct Obstruction in Patients Who Are Treated With Radioactive Iodine for Thyroid Cancer
Brief Title: Artificial Tears to Prevent Nasolacrimal Duct Obstruction in Patients Treated With Radioactive Iodine for Thyroid Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Rachel Sobel, Associate Professor of Ophthalmology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 230845
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Nasolacrimal Duct Obstruction; Thyroid Cancer
Keywords: Nasolacrimal Duct Obstruction; Artificial Tears; Thyroid Cancer
MeSH Terms: conditions — Lacrimal Duct Obstruction; Thyroid Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Artificial Tears) (Experimental): Participants in this arm will receive artificial tears to be administered in the 4 days immediately following radioactive iodine therapy. The schedule of administration will be as follows:
  Day 1 (day of radioactive iodine therapy): Every 15 minutes for 2 hours, then every 30 minutes for at least 4 hours or until bedtime at night Day 2: Once every 1 hour for 12 hours Day 3: Four times (approximately morning, lunch, dinner, and evening) Day 4: Two times (morning and evening)
  Interventions: Drug: Artificial Tears Methylcellulose
- No Intervention (No Artificial Tears) (No Intervention): Participants in this arm will not administer artificial tears in the 4 days immediately following radioactive iodine therapy.

INTERVENTIONS:
Drug: Artificial Tears Methylcellulose — Participants will self-administer the artificial tears according to the schedule.
  Arms: Experimental Arm (Artificial Tears)

SUMMARY:
The association of radioiodine therapy for the treatment of thyroid cancer with nasolacrimal duct obstruction has been well documented in the medical literature. Prior case reports have documented radioactive iodine detection in the tears of patients following radioiodine therapy. It is possible that radioactive uptake by the cells in the lacrimal sac and nasolacrimal duct lead to inflammation, fibrosis, and obstruction of the tear duct over time. A recent study has shown that the administration of artificial tears decreases the level of detectable radioiodine in the tears of patients undergoing radioiodine therapy for thyroid cancer. The purpose of this study will be to assess whether administering tears after radioactive iodine therapy for thyroid cancer decreases the incidence of nasolacrimal duct obstruction in the two years following radioactive iodine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Radio-iodine therapy for thyroid cancer
2. Radioiodine therapy ≥150 mCi
3. Age 18 or older

Exclusion Criteria:

1. Use of eye drops, other than artificial tears
2. History of periocular trauma with tear duct involvement/lacrimal gland trauma
3. History of lacrimal drainage disease: canaliculitis, dacryocystitis
4. Prior radiotherapy
5. Current or prior use of chemotherapy drugs (i.e. 5-fluorouracil, docetaxel)
6. Medical conditions that predispose to NLD stenosis (i.e. sarcoidosis, granulomatosis with polyangiitis, chronic lymphocytic leukemia)
7. Nasolacrimal duct obstruction at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-Radiotherapy Nasolacrimal Duct Obstruction (NLDO) | 2 years
  The rate of patients that developed NLDO after radioactive iodine therapy in each experimental group as determined by tear duct irrigation by an ophthalmologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No